CLINICAL TRIAL: NCT06187467
Title: Longitudinal Multimodal Profiling of Balance and Gait In Stroke Using EEG and Lower Limb Sensors: A Feasibility Study.
Brief Title: Longitudinal Multimodal Profiling of Balance and Gait In Stroke
Status: Recruiting | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Sponsor
Other Study IDs: DSRB 2023/00805
Record Dates: First submitted 2023-12-04; First posted 2024-01-02 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Electroencephalographic (EEG); Brain Computer Interfaces
MeSH Terms: conditions — Stroke | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Clinical and technological-aided assessments and questionnaires — Assessments and questionnaires to quantify cortical and motor activities using portable EEG and lower limb sensors during dynamic balance and gait activities.

SUMMARY:
Balance and gait recovery is a critical aspect of post-stroke motor rehabilitation. Researchers have effectively utilized EEG to investigate different aspects of lower limb motor control, however there are several technical challenges in the existing brain computer interface (BCI) motor profiling.

The study aims to test the EEG-BCI system to see if it's effective in understanding the balance and walking patterns of post-stroke populations.

DETAILED DESCRIPTION:
Brain Computer Interface represent a groundbreaking field at the crossroads of neuroscience and engineering, serving as a direct communication link between the human brain and computer system.

Despite advancements in BCI technology, the electrocortical oscillations during human walking remain relatively unexplored, providing an opportunity for pioneering investigations.

The research highlights the feasibility of using EEG to decode neural patterns associated with various functions and aims to contribute to existing knowledge by using advanced EEG-based techniques to predict balance and gait patterns with the ultimate goal of tailoring rehabilitation approaches to individual patient needs.

ELIGIBILITY:
Inclusion Criteria:

* First-ever clinical stroke (ischaemic or haemorrhagic) confirmed by admitting doctors brain imaging
* Age 21 to 85 years
* At least ≥ 30 days post-stroke
* Gait impairments related to stroke
* Functional ambulation category -6 levels (Mehrholz et al, 2007): FAC ≥ 4, i.e. able to ambulate independently on level surface but requires supervision to negotiate (e.g. stairs, inclines, non-level surfaces).
* Montreal Cognitive Assessment (MoCA) score > 21 (Nasreddine et al., 2005)
* Able to understand study instructions and requirements

Exclusion Criteria:

* Non-stroke related causes of gait impairment
* Medical conditions incompatible with research participation: uncontrolled medical illnesses (hypertension or diabetes, ischaemic heart disease, congestive heart failure, bronchial asthma, severe /untreated depression, agitation, end stage renal/liver/heart/lung failure, dialysis, unresolved cancers e.g.,), active seizures within 3 months
* Anticipated life expectancy of < 6 months
* On subcutaneous or oral anti-coagulation
* Local factors potentially worsened by gait training: joint and muscle pains
* Lower limb pain VAS >4/10, active lower limb fractures or arthritis, fixed leg contractures, severe peripheral vascular disease, organomegaly or aortic aneurysms
* Active unhealed skin wounds or inflammatory skin conditions over trunk and lower limbs,
* Severe visual impairment or visual neglect affecting navigation
* Known allergy to EEG gel (Recoverix)
* Presence of craniectomy skull defect
* Resident of nursing home or overseas country which may compromise attendance at research site
* Pregnant or lactating females

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
EEG Activities | Week 0 (baseline), 4 (1st follow-up assessment), 8 (last follow-up assessment)
  To record EEG and EOG data from 64-Ch ActiCap EEG cap and electrode
Goniometers | Week 0 (baseline), 4 (1st follow-up assessment), 8 (last follow-up assessment)
  7 sensors to measure 2-axis joint angles at bilateral Hip, Knee and Ankle

SECONDARY OUTCOMES:
Fugl Meyer Assessment for Lower Limbs | Week 0 (baseline), 4 (1st follow-up assessment), 8 (last follow-up assessment)
  Change in Fugl Meyer Motor Assessment score in the affected arm, minimum: 0, maximum: 66 with higher scores indicating greater levels of mobility function
Berg Balance Scale | Week 0 (baseline), 4 (1st follow-up assessment), 8 (last follow-up assessment)
  To assess functional balance
Modified Clinical Test for Sensory Interaction in Balance | Week 0 (baseline), 4 (1st follow-up assessment), 8 (last follow-up assessment)
  Assess complex sensory system to assist in determining which sensory system the individual relies upon (visual, somatosensory, vestibul)
10-metre Walk Test | Week 0 (baseline), 4 (1st follow-up assessment), 8 (last follow-up assessment)
  To assess walking speed over a short distance
6-minute Walk Test | Week 0 (baseline), 4 (1st follow-up assessment), 8 (last follow-up assessment)
  Determine the functional exercise capacity

CONTACTS AND LOCATIONS:
Overall Officials: Dr Wee Seng Kwee, Principal Investigator — Tan Tock Seng Hospital; Dr Karen Chua, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No